CLINICAL TRIAL: NCT03728673
Title: A Pilot Study Utilizing Escitalopram to Address Cognitive Dysfunction in Glioma Patients
Brief Title: A Study Utilizing Escitalopram in Glioma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0245-18-FB
Record Dates: First submitted 2018-10-19; First posted 2018-11-02 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2024-12

CONDITIONS: Glioma of Brain; Glioma
Keywords: serotonin selective reuptake inhibitor; cognition; escitalopram
MeSH Terms: conditions — Glioma | interventions — Escitalopram

STUDY DESIGN:
Intervention Model Description: Grade IV glioma or grade III astrocytoma participants will be treated with the selective serotonin reuptake inhibitor (SSRI) Escitalopram during a 17 week study period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Escitalopram (Experimental): In this open-label study, Escitalopram will be administered to all participants as 10 mg capsules to be taken by mouth daily for 90 days.
  Interventions: Drug: Escitalopram Oral Capsules

INTERVENTIONS:
Drug: Escitalopram Oral Capsules — Active capsules will contain 10 mg escitalopram oxalate.
  Other Names: escitalopram 10mg; Lexapro

SUMMARY:
Glioma is a cancer of glial cells, a class of tissue supporting neuronal function in the brain. As many as 85% of glioma patients experience cognitive impairment. This is not only from direct tumor involvement, but also from therapy such as cranial radiation and chemotherapy, which degrades neuronal function. There is evidence that serotonin selective reuptake inhibitors (SSRIs), such as escitalopram, improve cognition or prevent cognitive decline and may also improve outcomes critical to overall survival including functional independence, psychosocial stability, and quality of life. This pilot study will evaluate the effectiveness of the selective serotonin reuptake inhibitor (SSRI) escitalopram for treating cognitive impairment in newly diagnosed grade IV glioma over a 17 week treatment period.

DETAILED DESCRIPTION:
As many as 85% of patients with glioma, a cancer of glial cells, experience cognitive impairment. This is not only from direct tumor involvement, but also from therapy such as cranial radiation and chemotherapy, which degrades neuronal function. Commonly, impairments in visuospatial skills and executive function are seen. There is evidence that serotonin selective reuptake inhibitors (SSRIs) such as escitalopram improve modulation and function of resting state networks, contribute to neuroplastic changes in brain regions subserving these abilities, and provide general functional support to neuronal cells. In addition to either improving cognition or preventing cognitive decline, treatment with an SSRI may also improve outcomes critical to overall survival in this vulnerable population, including functional independence, psychosocial stability, and quality of life.

This study will characterize the degree of change in cognition/brain function in participants with grade IV glioma planning to undergo concurrent chemoradiation therapy followed by temozolomide and 17 weeks of treatment with an SSRI, escitalopram, and determine the degree of change in psychosocial function as assessed via ratings in mood and quality of life. The study hypothesis is that following treatment with escitalopram participants will experience improved cognitive and mood function over time.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven diagnosis of Grade IV glioma
* Newly diagnosed disease to receive chemotherapy and/or radiation
* Performance status Eastern Cooperative Oncology Group (ECOG) 0-2 or equivalent
* 19 years of age or older
* Life expectancy greater than 6 months
* Able to provide written informed consent for study participation
* Negative urine pregnancy test at enrollment for females of childbearing potential
* Female participants must be either post-menopausal (free from menses for 2 or more years), surgically sterilized, or willing to use two adequate barrier forms of contraception

Exclusion Criteria:

* Hemifield defects (obscures visual field necessary to participate in all tests)
* Inability to undergo MRI
* Severe renal impairment defined as Glomerular Filtration Rate (GFR) <30 mL/minute
* Screen positive for depression or anxiety
* Already taking an anti-depressant (SSRI or NSRI)
* Have problems tolerating past treatment with SSRI or NSRIs

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-03-06 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in Cognition | Baseline, 12-weeks and 17-weeks
  Changes in cognition will be measured using the NIH Toolbox neurocognitive assessments. The NIH Toolbox has excellent test / re-test reliability across composite domain scores r = .86 - .9263. It has also shown strong convergent (r = .78 - .9) and discriminant (r = .19 - .39) validities. It has been validated on groups of patients with Spinal Cord Injuries, Traumatic Brain Injury and Stroke. More recently a small group of patients diagnosed with diffuse glioma completed the NIH Toolkit Cognitive and Emotional batteries pre- and post-surgery. Results suggested good tolerance on the part of the patients and benefits of having a standardized battery that can be employed across sites.
  Paired t-test will be used to determine if the changes from baseline to the 17 week visit are significant. If assumptions for the paired t-test are not met, the non-parametric Wilcoxon sign rank test will be used instead.
Characterize the degree of change in cognition and brain function | Baseline, 12-weeks and 17-weeks
  Changes in cognition and brain function will be measured via Patient-Reported Outcome Measurement Information System (PROMIS) Neuro-QoL Item Bank v2.0 - Cognitive Function assessment completed at baseline, 12 weeks, and 17 weeks. A higher score on this measure indicate higher cognitive function.
  The change from baseline will be compared with the Wilcoxon sign rank test.
Change in Psycho-social Functions - PROMIS Neuro-QoL Item Bank v1.0 - Depression | Baseline, 12-weeks and 17-weeks
  The degree of change in psychosocial functions will be assessed via patient-reported ratings in mood and quality of life. The following assessments will be completed: PROMIS Neuro-QoL Item Bank v1.0 - Depression; PROMIS Neuro-QoL Item Bank v1.0 - Anxiety; PROMIS Neuro-QoL Item Bank v1.0 - Fatigue. Higher scores on these assessments indicate higher levels of the concept being assessed.
  The changes from baseline will be compared with the Wilcoxon sign rank test.
Change in Psycho-social Functions - PROMIS Neuro-QoL Item Bank v1.0 - Anxiety | Baseline, 12-weeks and 17-weeks
  The degree of change in psychosocial functions will be assessed via patient-reported ratings in mood and quality of life. The following assessments will be completed: PROMIS Neuro-QoL Item Bank v1.0 - Depression; PROMIS Neuro-QoL Item Bank v1.0 - Anxiety; PROMIS Neuro-QoL Item Bank v1.0 - Fatigue. Higher scores on these assessments indicate higher levels of the concept being assessed.
  The changes from baseline will be compared with the Wilcoxon sign rank test.
Change in Psycho-social Functions - PROMIS Neuro-QoL Item Bank v1.0 - Fatigue | Baseline, 12-weeks and 17-weeks
  The degree of change in psychosocial functions will be assessed via patient-reported ratings in mood and quality of life. The following assessments will be completed: PROMIS Neuro-QoL Item Bank v1.0 - Depression; PROMIS Neuro-QoL Item Bank v1.0 - Anxiety; PROMIS Neuro-QoL Item Bank v1.0 - Fatigue. Higher scores on these assessments indicate higher levels of the concept being assessed.
  The changes from baseline will be compared with the Wilcoxon sign rank test.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole A Shonka, MD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No